CLINICAL TRIAL: NCT07133022
Title: Effectiveness of Early Prone Positioning on Clinical Outcomes in Non-intubated Acute Respiratory Distress Syndrome (ARDS) Patients: A Quasi-experimental Study
Brief Title: Early Prone Positioning and Clinical Outcomes in Non-Intubated Acute Respiratory Distress Syndrome (ARDS) Patients
Acronym: EPP-ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loai Muawiah Zabin (Other)
Responsible Party: Sponsor-Investigator, Loai Muawiah Zabin, Assistant Professor, Faculty of Nursing, Arab American University (Palestine)
Organization: Arab American University (Palestine) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAUP-ARDS-2024; R-2024/B/84/N (Other: Institutional Review Board (IRB) at Arab American University-Palestine)
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Hypoxemia; Respiratory Failure; Non-Intubated Patients; Intensive Care Unit ICU
Keywords: Prone positioning; Non-invasive ventilation; Oxygenation; Intensive care unit; Early prone protocol; Low-resource settings; ARDS management; Clinical outcomes; Non-intubated ARDS; Critical care nursing; Quasi-experimental study; Palestine; Spontaneous breathing; ICU protocols
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the intervention group receiving early prone positioning or the control group receiving standard care. The study followed a quasi-experimental, non-randomized parallel assignment model.
Masking Description: None. Due to the physical nature of the intervention (prone positioning), blinding was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Prone Positioning Protocol (Experimental): Participants in this arm received early prone positioning as part of the study protocol. Patients were assisted into a prone position for 4 hours, with measurements taken at baseline, 2 hours, and 4 hours. The intervention was initiated soon after the Acute Respiratory Distress Syndrome (ARDS) diagnosis, according to clinical stability and eligibility. The procedure was supervised by trained Intensive Care Unit (ICU) nurses, with continuous monitoring for tolerance, oxygenation status, and safety.
  Interventions: Procedure: Early Prone Positioning Protocol
- Standard Care (Active Comparator): Participants in this arm received standard Intensive Care Unit (ICU) care without early implementation of prone positioning. Any use of prone positioning occurred at the discretion of the treating medical team and was not based on a standardized protocol. All other supportive treatments followed routine ICU protocols.
  Interventions: Other: Standard ICU Care

INTERVENTIONS:
Procedure: Early Prone Positioning Protocol — A structured protocol in which non-intubated patients with Acute Respiratory Distress Syndrome (ARDS) are positioned prone for 2-4 hours per session, multiple times per day, totaling approximately 8 hours daily for 5 consecutive days. Initiation begins within 24 hours of ARDS diagnosis. Administered by trained Intensive Care Unit (ICU) nurses under medical supervision.
  Other Names: Prone Positioning for ARDS
  Arms: Early Prone Positioning Protocol
Other: Standard ICU Care — Participants receive routine Intensive Care Unit (ICU) care for Acute Respiratory Distress Syndrome (ARDS) without the implementation of a structured early prone positioning protocol. Care is provided at the discretion of the treating physicians, following standard ICU management practices.
  Other Names: Usual ARDS Management
  Arms: Standard Care

SUMMARY:
This study aimed to evaluate the effectiveness of early prone positioning in improving clinical outcomes among non-intubated patients with Acute Respiratory Distress Syndrome (ARDS). Prone positioning, which involves placing patients on their stomachs, has been shown to improve outcomes in patients on mechanical ventilation. However, limited evidence exists for its use in non-intubated patients. The researchers conducted a quasi-experimental study at Jenin Governmental Hospital in Palestine, involving two groups: one received early prone positioning in addition to standard care, and the other received standard care alone. Key clinical outcomes included respiratory rate, oxygen saturation, need for intubation, length of Intensive Care Unit (ICU) stay, and mortality. This study adds to the growing evidence supporting non-invasive interventions for managing ARDS and may help inform future clinical guidelines in low-resource settings.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is a life-threatening condition characterized by rapid-onset respiratory failure, low blood oxygen levels (hypoxemia), and bilateral pulmonary infiltrates. While prone positioning has become an established part of care for intubated patients with moderate to severe ARDS, its role in non-intubated, spontaneously breathing patients remains underexplored, particularly in resource-limited settings.

This quasi-experimental study assessed the clinical effectiveness of early implementation of prone positioning in non-intubated ARDS patients in the Intensive Care Unit (ICU) of Jenin Governmental Hospital, Palestine. The study was conducted from January to April 2024. A total of 100 adult patients who met the Berlin definition of ARDS and did not require immediate intubation were enrolled and divided into two groups of 50: the intervention group received early prone positioning alongside standard medical care, while the control group received only standard care without prone positioning.

The primary clinical endpoints included changes in oxygen saturation (SpO₂), respiratory rate, need for mechanical ventilation, and length of ICU stay. Additional variables such as arterial blood gas (ABG) parameters, hemodynamic stability, and patient tolerance to prone positioning were monitored throughout the ICU admission. Patients were followed until ICU discharge or in-hospital mortality.

The early prone positioning protocol was implemented within 24 hours of ARDS diagnosis. Patients were assisted to maintain the prone position for multiple daily sessions, each lasting 2-4 hours, depending on tolerance and clinical stability. Standardized nursing assessments and physician evaluations were performed to monitor safety and efficacy.

Data were analyzed using appropriate statistical methods to compare outcomes between groups. Ethical approval was obtained from the Arab American University Institutional Review Board (IRB reference: R-2024/B/84/N). The study provides insight into the feasibility, safety, and potential clinical benefit of prone positioning as a low-cost, non-invasive intervention for managing ARDS in non-intubated patients, with implications for ICU protocols in low- and middle-income countries (LMICs).

ELIGIBILITY:
Inclusion Criteria:

* Awake patients diagnosed with Acute Respiratory Distress Syndrome (ARDS) according to established criteria.
* Eligible for prone positioning combined with non-invasive respiratory support.
* Willing and able to provide informed consent.
* Aged 18 years or older.
* Hemodynamically stable.
* Conscious, normal mental status, able to follow instructions, and capable of self-positioning.

Exclusion Criteria:

* Severe hemodynamic instability or other contraindications to prone positioning.
* Inability to provide consent or participate actively.
* Significant comorbidities that could confound outcomes.
* Impaired consciousness or inability to change position.
* Normal oxygen saturation without supplemental oxygen.
* Respiratory fatigue or patients receiving end-of-life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in arterial oxygenation (PaO₂ in mmHg) | Baseline, 2 hours, and 4 hours after intervention
  This outcome assesses the effect of early prone positioning on arterial oxygenation in non-intubated Acute Respiratory Distress Syndrome (ARDS) patients. The partial pressure of arterial oxygen (PaO₂) will be measured via arterial blood gas (ABG) analysis and compared between the intervention and control groups.

SECONDARY OUTCOMES:
Change in peripheral oxygen saturation (SpO₂ in %) | Baseline, 2 hours, and 4 hours after intervention
  Peripheral capillary oxygen saturation (SpO₂) will be measured using pulse oximetry to evaluate changes in oxygen saturation between intervention and control groups.
Change in respiratory rate (breaths/minute) | Baseline, 2 hours, and 4 hours after intervention
  Respiratory rate will be recorded by direct observation and counted per minute to assess improvement in breathing pattern.
Change in serum bicarbonate (HCO₃ in mmol/L) | Baseline, 2 hours, and 4 hours after intervention
  Bicarbonate (HCO₃) concentration will be obtained from arterial blood gas results to assess metabolic compensation.
Change in arterial carbon dioxide pressure (PaCO₂ in mmHg) | Baseline, 2 hours, and 4 hours after intervention
  Partial pressure of arterial carbon dioxide (PaCO₂) will be measured using arterial blood gas analysis to evaluate ventilatory status.
Change in blood pH | Baseline, 2 hours, and 4 hours after intervention
  Blood pH will be measured via arterial blood gas analysis to assess acid-base balance.
Incidence of complications | Baseline, 2 hours, and 4 hours after intervention
  Number of patients experiencing predefined complications (apnea, vomiting, discomfort, facial edema, decubitus ulcers) during ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Sajed Ghawadra, PhD, Study Chair — Arab American University (Palestine)
Locations (1):
- Jenin Governmental Hospital, Jenin, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional data protection policies, lack of dedicated infrastructure for secure data sharing, and the absence of participant consent for data sharing beyond the scope of the current study. Additionally, the study was conducted without external funding, which limits the capacity for data curation and repository access required for responsible sharing.